CLINICAL TRIAL: NCT03773185
Title: A Comparative Study of Brain Structure and Amyloid Load Between Cognitively Impaired Older People With or Without Diabetes Mellitus
Brief Title: A Comparative Study of Brain Structure and Amyloid Load in MCI Patients
Status: Withdrawn | Type: Observational
Why Stopped: Low recruitment rate
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Timothy Kwok, Professor, Chinese University of Hong Kong
Other Study IDs: 2018.454
Record Dates: First submitted 2018-11-30; First posted 2018-12-12 (Actual); Last update posted 2021-10-21 (Actual); Status verified 2021-10

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Older people with DM are at greater risk of cognitive decline than their counterparts with DM. Cognitive impairment in older people with DM may be associated with non-AD related brain atrophy and white matter disease. The investigators therefore propose to compare DM and non-DM older people with amnesic MCI in brian volumes, white matter disease and amyloid load.

30 older people with aMCI, 30 older people with aMCI and DM, age 65-85 will be recruited. They all will have amyloid PET scan and MRI brain scan.

ELIGIBILITY:
Inclusion Criteria:

* MCI patients

Exclusion Criteria:

* Patients with depression

Ages: 65 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: MCI patients with DM or without DM
Sampling Method: Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2018-12-15 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Amyloid load | Two years

CONTACTS AND LOCATIONS:
Overall Officials: Timothy Kwok, MD, Principal Investigator — Chinese University of Hong Kong
Locations (1):
- The Chinese University of Hong Kong, Hong Kong, Hong Kong